CLINICAL TRIAL: NCT04723056
Title: Zemedy - Evaluation of Zemedy, a Cognitive Behavioral Therapy-based Digital Therapeutic Application for the Treatment of Irritable Bowel Syndrome
Brief Title: Zemedy Application for Irritable Bowel Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of funding
Sponsor: Stanford University (Other)
Collaborators: Bold Health Inc. (Industry)
Responsible Party: Principal Investigator, Linda Nguyen, Clinical Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 59209
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Results first posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: IBS - Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Cognitive Behavioral Therapy; Self Help
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized trial comparing Zemedy CBT app vs. Treatment as usual
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Control Group (TAU only) (No Intervention): Treatment as Usual (TAU) for IBS patients are tailored to each individual's needs and may involve treatment such as: dietary modification, exercise, medication, and anti-diarrheal therapy.
- Experimental (TAU plus CBT) (Experimental): Subjects who are in the Experimental Group will receive 8 weeks of CBT from the Zemedy mobile application in addition to their treatment as usual (TAU).
  Interventions: Device: Use of Zemedy Application

INTERVENTIONS:
Device: Use of Zemedy Application — 8 weeks of CBT via the Zemedy Application.
  Arms: Experimental (TAU plus CBT)

SUMMARY:
The purpose of the study is investigate the effectiveness of Zemedy, a mobile application that enables the digital delivery of a CBT program to people with IBS.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is defined as having recurrent abdominal pain associated with defecation or a change of bowel habits. The pathophysiology of IBS can be looked through the biopsychosocial model of disease which is defined by the complex interplay between genetic, cultural, environmental, and psychosocial factors.

Treatment of IBS is multifaceted and ranges from exercise to dietary restrictions, however, psychological treatments to target the gut-brain axis such as cognitive-behavior therapy (CBT) have also been shown to be an effective therapy, and aims to address the psychological and environmental stressors that contribute to the symptoms. Therefore the purpose of the study is investigate the effectiveness of Zemedy, a mobile application that enables the digital delivery of a CBT program to people with IBS.

CBT has been shown to reduce the severity of intractable IBS symptoms by as much as 70%. The investigators hope to learn whether the Zemedy mobile application is effective in the reduction of IBS. This will be measured based on their IBS Symptom Severity Scores (SSS) at week 8 compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients >=18 years old.
2. Meet Rome IV criteria for IBS for at least 6 months. No restrictions on type of IBS.
3. English proficiency (in order to understand use of the application.
4. Patient must be on a stable regimen for IBS for at least 30 days.
5. Patients must own a smartphone (iOS or Android) in order to participate in the CBT application.

Exclusion Criteria:

1. Laboratory or imaging evidence of an alternative explanation of patient's symptoms.
2. Active gastrointestinal disease such as Crohn's disease, ulcerative colitis, history of complete colon resection, acute infection, or any disease that precludes participation in CBT application.
3. Patient already undergoing cognitive behavioral therapy.
4. Psychiatric hospitalization within 10 years.
5. Current or past diagnosis of a major mental illness such as schizophrenia, bipolar disorder, personality disorder or substance abuse.
6. Active (within the past 3 months) suicidal ideation.
7. Prisoners or other detained individuals.
8. Adults unable to consent.
9. Pregnant people.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Nguyen, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 21 participants signed informed consent; 18 were randomized to a study arm.
Groups:
- Experimental (TAU Plus CBT): Participants who are in the Experimental Group will receive 8 weeks of CBT from the Zemedy mobile application in addition to their treatment as usual (TAU).
Period: Overall Study
Arm/Group | Experimental (TAU Plus CBT) | Control Group (TAU Only)
Started | 9 | 9
Completed Week 8 Surveys | 7 | 8
Completed Week 24 Surveys | 7 | 8
Completed | 7 | 8
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental (TAU Plus CBT) | Control Group (TAU Only) | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Mean (Full Range); unit: years] | 36 [31 to 45] | 34 [29 to 38] | 35.5 [29 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 2 | 3 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9 | 7 | 16
  Non-white | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: IBS-SSS at 8 Weeks
Description: Change in IBS symptoms based on the change in IBS symptom severity score (IBS-SSS) score at week 8 compared to baseline. Score range: 0-500. Higher score corresponds to more severe symptoms (75-175 = mild, 176-300 - moderate; >300 = severe).
Time Frame: Baseline and at Week 8.
Population: Participants with data at the respective time point
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Experimental (TAU Plus CBT) | Control Group (TAU Only)
Number analyzed (Participants) | 9 | 9
score on a scale
  Baseline | 215 [174 to 268] | 171 [151 to 229]
  Week 8: number analyzed (Participants) | 7 | 8
  Week 8 | 126 [66 to 171] | 143.5 [119.5 to 197]
Statistical Analysis 1: Comparison: Experimental (TAU Plus CBT) vs Control Group (TAU Only); Between-group analysis at week 8; Test type: Other; p = 0.282, t-test, 2 sided — The a priori threshold for statistical significance was <0.05

2. Secondary Outcome: IBS-SSS at 24 Weeks
Description: Change in IBS symptoms based on the change in IBS symptom severity score (IBS-SSS) score at week 24 compared to baseline. Score range: 0-500. Higher score corresponds to more severe symptoms (75-175 = mild, 176-300 - moderate; >300 = severe).
Time Frame: Baseline and at Week 24
Population: Participants with data at the respective time point
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Experimental (TAU Plus CBT) | Control Group (TAU Only)
Number analyzed (Participants) | 9 | 9
score on a scale
  Baseline | 215 [174 to 268] | 171 [151 to 229]
  Week 24: number analyzed (Participants) | 7 | 8
  Week 24 | 134 [101 to 160] | 143.5 [119.5 to 197]
Statistical Analysis 1: Comparison: Experimental (TAU Plus CBT) vs Control Group (TAU Only); Between-group analysis at week 24; Test type: Other; p = 0.217, t-test, 2 sided — The a priori threshold for statistical significance was <0.05

3. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) - Depression Score
Description: Assesses mood measured by the total distress score (score range: 0 to 21; <7 normal, 8-14 borderline, 15 or >15, abnormal).
Time Frame: Baseline, week 8 and week 24
Population: Participants with data at the respective time point
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Experimental (TAU Plus CBT) | Control Group (TAU Only)
Number analyzed (Participants) | 9 | 9
score on a scale
  Baseline | 6 [4 to 7] | 2 [2 to 4]
  Week 8: number analyzed (Participants) | 7 | 8
  Week 8 | 7 [4 to 8] | 5 [3.5 to 7.5]
  Week 24: number analyzed (Participants) | 7 | 8
  Week 24 | 5 [3 to 6] | 1.5 [1 to 3]
Statistical Analysis 1: Comparison: Experimental (TAU Plus CBT) vs Control Group (TAU Only); Between-group analysis at week 8; Test type: Other; p = 0.462, t-test, 2 sided — The a priori threshold for statistical significance was <0.05
Statistical Analysis 2: Comparison: Experimental (TAU Plus CBT) vs Control Group (TAU Only); Between-group analysis at week 24; Test type: Other; p = 0.179, t-test, 2 sided — The a priori threshold for statistical significance was <0.05

4. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) - Anxiety Score
Description: as for outcome 3
Time Frame: Baseline, week 8 and week 24
Population: Participants with data at the respective time point
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Experimental (TAU Plus CBT) | Control Group (TAU Only)
Number analyzed (Participants) | 9 | 9
score on a scale
  Baseline | 10 [3 to 11] | 7 [5 to 10]
  Week 8: number analyzed (Participants) | 7 | 8
  Week 8 | 9 [8 to 10] | 8 [6 to 14.5]
  Week 24: number analyzed (Participants) | 7 | 8
  Week 24 | 8 [6 to 11] | 6.5 [3 to 10]
Statistical Analysis 1: Comparison: Experimental (TAU Plus CBT) vs Control Group (TAU Only); Between-group analysis at week 8; Test type: Other; p = .573, t-test, 2 sided — The a priori threshold for statistical significance was <0.05
Statistical Analysis 2: Comparison: Experimental (TAU Plus CBT) vs Control Group (TAU Only); Between-group analysis at week 24; Test type: Other; p = .606, t-test, 2 sided — The a priori threshold for statistical significance was <0.05

5. Secondary Outcome: Cohen Perceived Stress Questionnaire (PSQ)
Description: Measures degree situation's in one's life are seen as stressful (score range: 0 to 40; 0-13 = low stress, 14-26 = moderate stress, 27-40 = high stress)
Time Frame: baseline, 24 weeks
Population: Participants with data at the respective time point
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Experimental (TAU Plus CBT) | Control Group (TAU Only)
Number analyzed (Participants) | 9 | 9
score on a scale
  Baseline | 32 [27 to 34] | 21 [19 to 27]
  Week 24: number analyzed (Participants) | 7 | 8
  Week 24 | 29 [25 to 35] | 22 [18 to 28]
Statistical Analysis 1: Comparison: Experimental (TAU Plus CBT) vs Control Group (TAU Only); Between-group analysis at week 24; Test type: Other; p = .181, t-test, 2 sided — The a priori threshold for statistical significance was <0.05

6. Secondary Outcome: Work and Social Adjustment Scale (WSAS)
Description: Measures the effect of IBS on ability to work and manage at home, participate in social and private leisure activities and maintain relationships. Score range: 0 to 40 (<10 subclinical/mild, 10-20 significant, >20 severe).
Time Frame: Baseline, week 24
Population: Participants with data at the respective time point
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Experimental (TAU Plus CBT) | Control Group (TAU Only)
Number analyzed (Participants) | 9 | 9
score on a scale
  Baseline | 14 [7 to 16] | 13 [11 to 18]
  Week 24: number analyzed (Participants) | 7 | 8
  Week 24 | 9 [6 to 14] | 14.5 [9 to 16]
Statistical Analysis 1: Comparison: Experimental (TAU Plus CBT) vs Control Group (TAU Only); Between-group analysis at week 24; Test type: Other; p = .407, t-test, 2 sided — The a priori threshold for statistical significance was <0.05

7. Secondary Outcome: Subject's Global Assessment of Relief (SGA)
Description: Assesses global symptoms relief asking the question, "Overall, how do you feel?". Score range: -2 (no pain) to +2 (severe pain/discomfort).
Time Frame: Baseline, Week 24
Population: Participants with data at the respective time point
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Experimental (TAU Plus CBT) | Control Group (TAU Only)
Number analyzed (Participants) | 9 | 9
score on a scale
  Baseline | 0 [-1 to 0] | 1 [0 to 1]
  Week 24: number analyzed (Participants) | 7 | 8
  Week 24 | 0 [-1 to 1] | 1.5 [0 to 2]
Statistical Analysis 1: Comparison: Experimental (TAU Plus CBT) vs Control Group (TAU Only); Between-group analysis at week 24; Test type: Other; p = .643, t-test, 2 sided — The a priori threshold for statistical significance was <0.05

8. Secondary Outcome: Work Productivity and Activity Impairment (WPAI) Questionnaire
Description: Assesses work productivity based on percentage of work days taken off due to health
Time Frame: Baseline, 8 weeks, 24 weeks
Population: Participants with data at the respective time point
Measure: Mean (Standard Deviation); unit: percentage of work time missed
Arm/Group | Experimental (TAU Plus CBT) | Control Group (TAU Only)
Number analyzed (Participants) | 9 | 9
percentage of work time missed
  Baseline | 9.59 (6.06) | 3.57 (4.65)
  Week 8: number analyzed (Participants) | 7 | 8
  Week 8 | 2.6 (4.1) | 1.5 (3.3)
  Week 24: number analyzed (Participants) | 7 | 8
  Week 24 | 1.4 (1.8) | 0.96 (1.9)
Statistical Analysis 1: Comparison: Experimental (TAU Plus CBT) vs Control Group (TAU Only); Between-group analysis at week 8; Test type: Other; p = .625, t-test, 2 sided — The a priori threshold for statistical significance was <0.05
Statistical Analysis 2: Comparison: Experimental (TAU Plus CBT) vs Control Group (TAU Only); Between-group analysis at week 24; Test type: Other; p = .707, t-test, 2 sided — The a priori threshold for statistical significance was <0.05

9. Secondary Outcome: Number of Participants Who Had an Urgent Care, Emergency Department, or Physician Appointment Due to IBS
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental (TAU Plus CBT) | Control Group (TAU Only)
Number analyzed (Participants) | 9 | 9
Participants
  Urgent care | 0 | 0
  Emergency Department | 1 | 0
  Physician appointment | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Experimental (TAU Plus CBT) | Control Group (TAU Only)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 1/9 | 0/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (TAU Plus CBT) (N=9) | Control Group (TAU Only) (N=9)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 — Unrelated to treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT04723056/Prot_SAP_000.pdf